CLINICAL TRIAL: NCT03336099
Title: Evolution of Clinical State of Patients With Rheumatic Disease on Lower Limbs or Rachis, 6 Months After Spa Treatment
Brief Title: Assessment of the Effect of Spa Treatment on the Functional Severity of Arthrosis
Acronym: VALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Le Syndicat Intercommunal pour le Thermalisme et l'Environnement (Other)
Collaborators: Floralis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 2.0
Record Dates: First submitted 2017-04-24; First posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Osteoarthritis, Knee; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spa Treatment (Experimental): Bicarbonate and sulfurated water cares in Vals-les-Bains thermal cure center, massage, cataplasm.
  Interventions: Other: Spa Treatment

INTERVENTIONS:
Other: Spa Treatment — * Bath with immersion shower
  * Overall shower, penetrating shower
  * Multiple local application cataplasm
  * Single local application cataplasm
  * Inhalation or collective steam bath
  * Individual physiotherapy technique

SUMMARY:
Assessment of the effect of spa treatment on the functional severity of arthrosis.

Official title: Evolution of clinical state of patients with rheumatic disease on lower limbs or rachis, 6 months after spa treatment.

Primary outcome measure:

* Measuring the effect of spa treatment on functional severity of arthrosis

  * Proportion of patients with a WOMAC score augmented by 9 or more, 6 months after enrollment (minimal clinically important difference)

Secondary outcome measures

* Quantitative evaluation of pain

  * Comparison of mean Visual Analogue Scale (VAS) pain scale between enrollment and 6 months after
* Quantitative evaluation of WOMAC

  * Comparison of mean WOMAC between enrollment and 6 months after
* Impact of spa treatment on the patient's metabolism

  * Height and Weight (BMI calculation)
  * Blood pressure
  * Heart rate
* Quality of life

  * 36-Item Short Form (SF36) at enrollment, 3 months and 6 months
  * EuroQol 5 Dimensions (EQ5D) questionnaire at enrollment, 3 months and 6 months
* Opinion of doctor and patient

  * Semi-quantitative scale collected at enrollment, 3 months and 6 months
* Treatment follow-up
* Self-evaluation of pain

  * Self-evaluation of pain with VAS pain scale every 6 week

DETAILED DESCRIPTION:
Arthrosis and rheumatic diseases on the whole consist in a huge and frequent public health problem, with consequences notably including the well-known pain phenomena.

Spa treatments are part of the mainstream therapeutic arsenal of non-medical treatments proposed to this kind of patients.

A recent French study estimated the direct cost of arthrosis in France to 1.6 billion euros in 2002. Half of it was attributable to hospital expenses (800 million euros). Arthrosis required 13 million consultations and drug expenses amounting to 570 million euros. These expenses were increased by 156% compared to 1993 due to the raise of the number of treated patients (+54%) and the cost for each patient (+2.5% per year). This study concerned patients with arthrosis on the lower limbs, with an significant portion of these expenses attributable to the disease.

Different thermal clinical trials of good quality have led to the recognition of spa in the treatment of chronic low back pain.

Several controlled and randomized prospective trials already evaluated the effect of spa treatment for the other main indications claimed by crenotherapy in rheumatology : chronic low back pain, coxarthrosis, hand arthrosis, fibromyalgia, rheumatoid polyarthritis, psoriatic arthritis, chronic cervicalgia.

The THERMARTHROSE study by Forestier has demonstrated the efficacy of spa treatment as a rheumatologic indication for gonarthrosis on WOMAC and VAS pain scale. Following the model of this study, the sponsor chose to use the WOMAC as the primary endpoint for the VALS study.

It has been developed by Bellamy in 1988, and it is a functional index aimed on the locomotor system.

Nowadays, the WOMAC is more used than the Lequesne index because it has better internal consistency reliability. However, complementary validation efforts were necessary to calculate the minimal clinically important difference whereas the pertinence of the Lequesne index is immediately perceptible, being purely qualitative.

With studies in thermal environment, spa treatment is a composite entity including the effect of water itself, but also kinesiotherapy, rest, education… The spa of Vals-les-Bains wishes to obtain a new therapeutic orientation: the rheumatologic orientation. According to the recommendations of the Academy of Medicine, a prolonged observation of a cohort with repeated measures is required for any spa wishing to acquire the accreditation for a new orientation.

Toward this goal, the sponsor wish to undertake a prospective study with repeated measures in order to analyze the evolution at 6 month of the clinical state of patients with a rheumatologic disease on the lower limbs or the rachis and taken over for spa treatment at Vals-les-Bains. Since rheumatologic treatments at Vals-les-Bains are not covered by the health insurance, they will not be billed to the patients

ELIGIBILITY:
Inclusion Criteria:

* Patient with arthrosis or other rheumatic disease, located on the lower limbs or the rachis
* Rheumatic indication for spa treatment
* Diminution of mobility
* Affiliation to the French social security system or equivalent
* Available for a 6-months follow-up and an 18-days spa treatment

Exclusion Criteria:

* Pregnancy, parturient or breast feeding
* Psychiatric illness or social situation that would preclude study compliance
* Contraindication to spa treatment
* Predictable intolerance to thermal treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
Measuring the effect of spa treatment on functional severity of arthrosis | 6 months
  Proportion of patients with a WOMAC score augmented by 9 or more, at 6 months compared to baseline (minimal clinically important difference)

SECONDARY OUTCOMES:
Quantitative evaluation of pain | at baseline, 3 and 6 months
  Comparison of mean VAS pain scale between baseline, 3 and 6 months
Quantitative evaluation of WOMAC | at baseline, 3 and 6 months
  Comparison of mean WOMAC between baseline, 3 months and 6 months
Patient's BMI | at baseline, 3 and 6 months
  weight and height will be combined to report BMI in kg/m2
Quality of life | at baseline, 3 and 6 months
  SF36 questionnaire at baseline, 3 and 6 months
Quality of life | at baseline, 3 and 6 months
  EQ5D questionnaire at baseline, 3 and 6 months
Opinion of doctor and patient | at baseline, 3 and 6 months
  Semi-quantitative scale collected at baseline, 3 and 6 months
Number of treatments prescribed | at baseline, 3 and 6 months
  Type of treatments prescribed at baseline, 3 and 6 months will be collected
Changes in treatments prescribed | at baseline, 3 and 6 months
  changes in treatments prescribed at baseline, 3 and 6 months will be collected
Treatments duration | at baseline, 3 and 6 months
  Duration of treatments prescribed at baseline, 3 and 6 months will be collected
Self-evaluation of pain | at baseline, 1.5, 3, 4.5 and 6 months
  Self-evaluation of pain with VAS pain scale at baseline, 1.5, 3, 4.5 and 6 months
patient examination | at baseline, 3 and 6 months
  heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic BACONNIER, Principal Investigator — Ardèche Méridionale Hospital
Locations (1):
- Thermes de Vals Les Bains, Vals-les-Bains, Ardèche, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buskila D, Abu-Shakra M, Neumann L, Odes L, Shneider E, Flusser D, Sukenik S. Balneotherapy for fibromyalgia at the Dead Sea. Rheumatol Int. 2001 Apr;20(3):105-8. doi: 10.1007/s002960000085. PMID 11354556
- [Background] Constant F, Collin JF, Guillemin F, Boulange M. Effectiveness of spa therapy in chronic low back pain: a randomized clinical trial. J Rheumatol. 1995 Jul;22(7):1315-20. PMID 7562765
- [Background] Elkayam O, Ophir J, Brener S, Paran D, Wigler I, Efron D, Even-Paz Z, Politi Y, Yaron M. Immediate and delayed effects of treatment at the Dead Sea in patients with psoriatic arthritis. Rheumatol Int. 2000;19(3):77-82. doi: 10.1007/s002960050107. PMID 10776684
- [Background] Franke A, Reiner L, Pratzel HG, Franke T, Resch KL. Long-term efficacy of radon spa therapy in rheumatoid arthritis--a randomized, sham-controlled study and follow-up. Rheumatology (Oxford). 2000 Aug;39(8):894-902. doi: 10.1093/rheumatology/39.8.894. PMID 10952746
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- [Background] Konrad K, Tatrai T, Hunka A, Vereckei E, Korondi I. Controlled trial of balneotherapy in treatment of low back pain. Ann Rheum Dis. 1992 Jun;51(6):820-2. doi: 10.1136/ard.51.6.820. PMID 1535495
- [Background] Leplege A, Ecosse E, Verdier A, Perneger TV. The French SF-36 Health Survey: translation, cultural adaptation and preliminary psychometric evaluation. J Clin Epidemiol. 1998 Nov;51(11):1013-23. doi: 10.1016/s0895-4356(98)00093-6. PMID 9817119
- [Background] Neumann L, Sukenik S, Bolotin A, Abu-Shakra M, Amir M, Flusser D, Buskila D. The effect of balneotherapy at the Dead Sea on the quality of life of patients with fibromyalgia syndrome. Clin Rheumatol. 2001;20(1):15-9. doi: 10.1007/s100670170097. PMID 11254234
- [Background] Tubach F, Ravaud P, Baron G, Falissard B, Logeart I, Bellamy N, Bombardier C, Felson D, Hochberg M, van der Heijde D, Dougados M. Evaluation of clinically relevant states in patient reported outcomes in knee and hip osteoarthritis: the patient acceptable symptom state. Ann Rheum Dis. 2005 Jan;64(1):34-7. doi: 10.1136/ard.2004.023028. Epub 2004 May 6. PMID 15130902
- [Background] van Tubergen A, Landewe R, van der Heijde D, Hidding A, Wolter N, Asscher M, Falkenbach A, Genth E, The HG, van der Linden S. Combined spa-exercise therapy is effective in patients with ankylosing spondylitis: a randomized controlled trial. Arthritis Rheum. 2001 Oct;45(5):430-8. doi: 10.1002/1529-0131(200110)45:53.0.co;2-f. PMID 11642642
- [Background] Van Tubergen A, Boonen A, Landewe R, Rutten-Van Molken M, Van Der Heijde D, Hidding A, Van Der Linden S. Cost effectiveness of combined spa-exercise therapy in ankylosing spondylitis: a randomized controlled trial. Arthritis Rheum. 2002 Oct 15;47(5):459-67. doi: 10.1002/art.10658. PMID 12382292
- [Background] Verhagen AP, de Vet HC, de Bie RA, Kessels AG, Boers M, Knipschild PG. Balneotherapy for rheumatoid arthritis and osteoarthritis. Cochrane Database Syst Rev. 2000;(2):CD000518. doi: 10.1002/14651858.CD000518. PMID 10796385
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Forestier R, Desfour H, Tessier JM, Francon A, Foote AM, Genty C, Rolland C, Roques CF, Bosson JL. Spa therapy in the treatment of knee osteoarthritis: a large randomised multicentre trial. Ann Rheum Dis. 2010 Apr;69(4):660-5. doi: 10.1136/ard.2009.113209. Epub 2009 Sep 3. PMID 19734131